CLINICAL TRIAL: NCT02244034
Title: Incidence and Risk Factors of Postoperative Hypothermia in Patients With Cardiopulmonary Bypass.
Brief Title: Incidence and Risk Factors of Postoperative Hypothermia in Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Chaowanan Khamtuikrua, instructor, Mahidol University
Other Study IDs: SI002
Record Dates: First submitted 2014-09-15; First posted 2014-09-18 (Estimated); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Postoperative Hypothermia in Patients With Cardiopulmonary Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 760 patients who underwent open cardiac and/or thoracic aortic surgery using CPB
  Interventions: Procedure: hypothermia

INTERVENTIONS:
Procedure: hypothermia

SUMMARY:
Background: Postoperative hypothermia may result in relevant complications such as adverse cardiovascular events, wound infection, and coagulopathy with consecutive blood loss. Patients with open cardiac surgery using cardiopulmonary bypass are particular at risk for hypothermia. The study of Karalapillai and coworkers, analyzing a huge database incl. 43,158 patients with CPB, revealed 66% of them experiencing postoperative hypothermia during the first 24 hours and 0.3% longer than that. During cardiac surgery great parts of body surface including wound surface are exposed. Many of these patients receive large amounts of infusions and transfusions, and undergo hemodilution during CPB, which may additionally contribute to development of hypothermia.

Objective of the planned study is to find out incidence and duration of postoperative hypothermia and also risk factors for hypothermia in cardiac patients. Further objective is the incidence of postoperative complications and its relation to postoperative core temperature.

Methods: A retrospective chart review 780 patients who had been underwent cardiac surgery with CPB Included are patients ≥ 18 years old. Excluded are patients with preoperative hyperthermia (> 37.8 °C) and hypothermia (> 36 °C).

The following parameters will be recorded: temperature is measured at ICU after arrived and after 6 hours which is primary outcome, biometric data include age, sex, body weight, height, ASA physical status, surgical procedure includes emergency cases, anesthetic and surgical (bypass-) times, infusion/transfusion-regimen, blood loss and urine output, coolest temperature during bypass, method of temperature protection, and the outcome of operation .

All data will be described in number and percent and Pearson chi-square method will be used for analyze correlation between hypothermia and risk factor . P-value <0.05 will be defined to significant.

ELIGIBILITY:
Inclusion Criteria:

* patients ≥ 18 years old

Exclusion Criteria:

* patients with preoperative hyperthermia (> 37.8 °C) and hypothermia (< 36 °C).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who had been underwent cardiac surgery with CPB during 2012-2013
Sampling Method: Non-Probability Sample
Enrollment: 760 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2013-12-31 (Actual)

PRIMARY OUTCOMES:
incidence of postoperative hypothermia in patients with cardiopulmonary bypass. | 24 hours
  Upon arrival at the Cardiac Surgical Intensive Care Unit (CSICU), body temperature was measured using an infrared tympanic membrane thermometer. Postoperative hypothermia, which was defined as the body temperature < 36 degrees C upon arrival at the CSICU.

SECONDARY OUTCOMES:
predictors of postoperative hypothermia in patients with cardiopulmonary bypass. | 24 hours
  Predictors such as age, sex, body surface area, emergency surgery, time of operation, time of cardiopulmonary bypass time, fluid and blood component administer will be analyze.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine Siriraj hospital, Bangkok, Thailand